CLINICAL TRIAL: NCT02684799
Title: A Phase 1, Single and Multiple-Dose, Open-Label Study in Healthy Subjects to Assess the Effect of the Acid Reducing Agents, Omeprazole (OME) and Famotidine (FAM), on the Pharmacokinetics (PK) of Cenicriviroc Mesylate (CVC)
Brief Title: Pharmacokinetic and Safety Study of Cenicriviroc and Acid Reducing Agents When Dosed Alone or in Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 652-123
Record Dates: First submitted 2016-02-03; First posted 2016-02-18 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — cenicriviroc; Omeprazole; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1 Group 1 (Cenicriviroc) (Experimental): Part 1 Group 1 (12 subjects) will receive CVC 150 mg on Days 1, 7 and 13.
  Interventions: Drug: Cenicriviroc
- Part 1 Group 1 (Omeprazole) (Active Comparator): Part 1 Group 1 (12 subjects) will receive Omeprazole 20 mg from Days 2-7, and Omeprazole 40 mg from Days 8-13.
  Interventions: Drug: Omeprazole
- Part 1 Group 2 (Cenicriviroc) (Experimental): Part 1 Group 2 (12 subjects) will receive CVC 150 mg on Days 1, 5, 9 and 13.
  Interventions: Drug: Cenicriviroc
- Part 1 Group 2 (Famotidine) (Active Comparator): Part 1 Group 2 (12 subjects) will receive Famotidine 40 mg on Days 5, 9 and 13.
  Interventions: Drug: Famotidine
- Part 2 (Cenicriviroc) (Experimental): Part 2 (24 subjects) will receive Cenicriviroc from Days 1-10 and Days 11-20.
  Interventions: Drug: Cenicriviroc
- Part 2 (Omeprazole) (Active Comparator): Part 2 (24 subjects) will receive Omeprazole from Days 11-20.
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Cenicriviroc
  Other Names: Cenicriviroc 150 mg
  Arms: Part 1 Group 1 (Cenicriviroc); Part 1 Group 2 (Cenicriviroc); Part 2 (Cenicriviroc)
Drug: Omeprazole
  Other Names: Omeprazole 20 mg; Omeprazole 40 mg
  Arms: Part 1 Group 1 (Omeprazole); Part 2 (Omeprazole)
Drug: Famotidine
  Other Names: Famotidine 40 mg
  Arms: Part 1 Group 2 (Famotidine)

SUMMARY:
This is a Phase 1, Single and Multiple-Dose, Open-Label Study in Healthy Subjects to Assess the Effect of the Acid Reducing Agents, Omeprazole and Famotidine, on the PK of CVC

ELIGIBILITY:
Inclusion Criteria:

* Be informed of the nature of the study and have provided written informed voluntary consent.
* Have a BMI ≥ 18.0 and ≤ 35.0 kg/m2.
* Be in good general health with no clinically relevant abnormalities based on medical history, physical examination, clinical laboratory evaluations (clinical chemistry, hematology, urinalysis), and 12-lead ECG that, in the opinion of the Investigator, would affect subject safety.
* Be able to communicate effectively with the Investigator and other study center personnel and agree to comply with the study procedures and restrictions.

Exclusion Criteria:

* Any disease or condition that might affect drug absorption, metabolism, or excretion, or clinically significant cardiovascular, hematological, renal, hepatic, pulmonary, endocrine, gastrointestinal, immunological, dermatological, neurological, or psychiatric disease, as determined by the Investigator and, if necessary, the Sponsor's Medical Monitor.
* History of stomach or intestinal surgery, except for fully healed appendectomy and/or cholecystectomy which will be allowed.
* Clinically significant illness or clinically significant surgery within 4 weeks before the administration of study medication.
* History of GERD, heartburn, or nausea more than once a month, or any similar symptoms requiring the regular use of antacids, or any use of H2 histamine blockers or proton-pump inhibitors over the past 3 months.
* History of achlorhydria, pernicious anemia, or peptic ulcers over the past 6 months.
* Have a positive Helicobacter pylori urea breath test.
* Known or suspected hypersensitivity or allergic reaction to any of the components of CVC, OME or FAM tablets.
* History of malignancy, with the exception of cured basal cell or squamous cell carcinoma of the skin.
* If female, is pregnant or breast feeding, or has a positive pregnancy test result prior to the first dose of study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2016-04-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Assessment of CVC, as measured by maximum plasma concentration (Cmax) | Days 1, 7, and 13 for Part 1 Group 1. Days 1, 5, 9, and 13 for Part 1 Group 2.
Pharmacokinetic Assessment of CVC, as measured by minimum plasma concentration (Cmin) | Days 1, 7, and 13 for Part 1 Group 1. Days 1, 5, 9, and 13 for Part 1 Group 2.
Pharmacokinetic Assessment of CVC, as measured by area under the plasma concentration-time curve (AUC) | Days 1, 7, and 13 for Part 1 Group 1. Days 1, 5, 9, and 13 for Part 1 Group 2.

SECONDARY OUTCOMES:
Evaluation of Adverse Events | 23 days
  Evaluate adverse events
Changes from Baseline in Clinical Laboratory Tests | Baseline and 23 days
  Evaluate changes from baseline in clinical laboratory tests including serum chemistry, hematology and urinalysis
Changes from Baseline in 12-lead ECGs | Baseline and 23 days
  Evaluate changes from baseline in 12-lead ECGs
Changes from Baseline in Vital Signs | Baseline and 23 days
  Evaluate changes from baseline in vital signs, including blood pressure and pulse rate
Changes from Baseline in Physical Examinations | Baseline and 23 days
  Evaluate changes from baseline in physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Star Seyedkazemi, PharmD, Study Director — Tobira Therapeutics, Inc.
Locations (1):
- SeaView Research, Inc., Miami, Florida, United States